CLINICAL TRIAL: NCT01427140
Title: Metabolic Consequences of Moderate Weight Gain - Role of Dietary Fat Composition (LIPOGAIN): a Randomized Double-Blind Controlled Study
Brief Title: Metabolic Consequences of Moderate Weight Gain - Role of Dietary Fat Composition (LIPOGAIN)
Acronym: LIPOGAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SLS-2011-LPG
Record Dates: First submitted 2011-08-19; First posted 2011-09-01 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Liver fat; Polyunsaturated fatty acids (PUFA); Saturated fatty acids (SFA); Weight gain; Overfeed; Dietary fatty acids; Palm oil; Sunflower oil
MeSH Terms: conditions — Fatty Liver; Weight Gain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saturated fatty acid group (Active Comparator): Addition of saturated fatty acids to the diet inte the form of pastries
  Interventions: Other: Saturated fatty acid group
- Polyunsaturated fatty acid group (Active Comparator): Addition of polyunsaturated fatty acids to the diet in the form of pastries
  Interventions: Other: Polyunsaturated fatty acid group

INTERVENTIONS:
Other: Polyunsaturated fatty acid group — Addition of polyunsaturated fatty acids to the diet in the form of pastries
  Arms: Polyunsaturated fatty acid group
Other: Saturated fatty acid group — Addition of saturated fatty acids to the diet in the form of pastries
  Arms: Saturated fatty acid group

SUMMARY:
The purpose of this study is to investigate the metabolic consequences of a moderate weight gain and if the type of dietary fat (saturated versus polyunsaturated) can modify the effects in young healthy adults. Hypothesis: the type of dietary fat can modify the effects of weight gain.

DETAILED DESCRIPTION:
Specific goals:

* Investigate if dietary fat composition influences liver fat accumulation and metabolic risk factors in response to moderate weight gain
* Investigate if polyunsaturated fat (PUFA) in the diet could counteract any unfavorable metabolic changes that are expected to accompany moderate weight gain
* Investigate effects of weight gain and dietary fat composition on markers of vascular health

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* Body Mass Index 18-27

Exclusion Criteria:

* Liver disease,
* Coronary heart disease,
* Diabetes mellitus,
* Malignant diseases,
* Alcohol or drug abuse,
* Magnetic Resonance-incompatibility,
* Abnormal clinical chemistry,
* Use of drugs that significantly effects energy metabolism,
* Heavy exercise,
* Pregnancy or lactation,
* Allergy of gluten, egg or milk protein

Ages: 20 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Hepatic steatosis by magnetic resonance tomography (MRT) | 6 weeks

SECONDARY OUTCOMES:
high density lipoprotein (HDL) | 6 weeks
low density lipoprotein (LDL) | 6 weeks
Insulin | 6 weeks
Glucose | 6 weeks
Triglycerides | 6 weeks
Cholesterol | 6 weeks
Apolipoprotein B (ApoB) | 6 weeks
Apolipoprotein A1 (ApoA1) | 6 weeks
Aspartate aminotransferase (ASAT) | 6 weeks
Alanine aminotransferase (ALAT) | 6 weeks
Gamma glutamyl transpeptidase (GGT) | 6 weeks
Homeostasis model of assessment insulin resistance (HOMA-IR) | 6 weeks
C-reactive protein (CRP) | 6 weeks
Proinsulin | 6 weeks
Endostatin | 6 weeks
Pentraxin-3 (PTX-3) | 6 weeks
Endothelin-1 (ET-1) | 6 weeks
E-selectin | 6 weeks
Cathepsin-S | 6 weeks
Cystatin C | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Risérus, Ass. professor, Principal Investigator — Clinical Nutrition and Metabolism, Dept. of Public Health and Caring Sciences, Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala Science Park, Uppsala, Sweden

REFERENCES:
- [Derived] Rosqvist F, Orho-Melander M, Kullberg J, Iggman D, Johansson HE, Cedernaes J, Ahlstrom H, Riserus U. Abdominal Fat and Metabolic Health Markers but Not PNPLA3 Genotype Predicts Liver Fat Accumulation in Response to Excess Intake of Energy and Saturated Fat in Healthy Individuals. Front Nutr. 2020 Dec 3;7:606004. doi: 10.3389/fnut.2020.606004. eCollection 2020. PMID 33344496
- [Derived] Perfilyev A, Dahlman I, Gillberg L, Rosqvist F, Iggman D, Volkov P, Nilsson E, Riserus U, Ling C. Impact of polyunsaturated and saturated fat overfeeding on the DNA-methylation pattern in human adipose tissue: a randomized controlled trial. Am J Clin Nutr. 2017 Apr;105(4):991-1000. doi: 10.3945/ajcn.116.143164. Epub 2017 Mar 8. PMID 28275132
- [Derived] Iggman D, Rosqvist F, Larsson A, Arnlov J, Beckman L, Rudling M, Riserus U. Role of dietary fats in modulating cardiometabolic risk during moderate weight gain: a randomized double-blind overfeeding trial (LIPOGAIN study). J Am Heart Assoc. 2014 Oct 15;3(5):e001095. doi: 10.1161/JAHA.114.001095. PMID 25319187